CLINICAL TRIAL: NCT05004025
Title: Single Arm Trial of Tumor-Treating Fields in Combination With Nivolumab and Ipilimumab in Metastatic Uveal Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTFields-UM
Record Dates: First submitted 2021-06-16; First posted 2021-08-13 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Tumor-Treating Fields in Combination with Immunotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TTF Plus Chemotherapy (Experimental): Novacure Optune with Opdivo and Yervoy
  Interventions: Device: Novocure Optune; Drug: Opdivo; Drug: Yervoy

INTERVENTIONS:
Device: Novocure Optune — Novacure Optune with Opdivo and Yervoy
Drug: Opdivo — Novacure Optune with Opdivo and Yervoy
  Other Names: Nivolumab
Drug: Yervoy — Novacure Optune with Opdivo and Yervoy
  Other Names: Ipilimumab

SUMMARY:
Tumor Treating Fields targeted to liver metastases may improve outcomes for patients with metastatic uveal melanoma treated with immune checkpoint inhibitors.

DETAILED DESCRIPTION:
Uveal melanoma is the most common ocular malignancy for adults and despite effective therapies, roughly 50% of patients will develop metastatic disease. Currently there is no therapy to improve the prognosis of patients with metastatic disease and these patients are usually treated with regimens used for cutaneous melanoma. Tumor Treating Fields is a new type of anti-cancer therapy approved by the FDA for use in glioblastoma multiforme and mesothelioma. TTF has been shown to activate the STING pathway leading to increased levels of dendritic cells in regional lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has histologically or cytologically confirmed metastatic uveal melanoma with predominant liver involvement
2. Age 18 years or older and willing and able to provide informed consent
3. WOCBP must have a negative serum pregnancy test documented with 72 hours of first administration of drug
4. Sexually active and WOCBP, patient and partner must agree to use adequate contraception
5. Normal organ and marrow function
6. ECOG 0-1
7. Life expectancy of 3 months or greater

Exclusion Criteria:

1. History of previous grade 3, life threatening immune related adverse event (irAE) from prior checkpoint inhibitor therapy
2. Prior treatment with anti cytotoxic T-Lymphocyte-Associated protein 4 (CTLA-4) therapy within 90 days of C1D1 of study treatment
3. Prior anti-cancer therapy (systemic, regional or radiation) within 2 weeks of C1D1 of study treatment
4. AEs from prior anticancer therapies that have not resolved to grade 1 or less, other than endocrine related irAEs for which patients are on appropriate replacement therapy (ie hypothyroidism, adrenal insufficiency, type 1 diabetes)
5. History of or active autoimmune disease requiring systemic corticosteroid or immunosuppressive therapy. (Patients who have limited autoimmune disease not requiring systemic therapy or autoimmune disease that is unlikely to recur, such as ulcerative colitis s/p colectomy, will be allowed to enroll.)
6. Serious medical risk factors involving any of the major organ systems such that the Investigator considers it unsafe for the patient to receive an experimental research drug.
7. Patient is unwilling or unable to comply with study procedures
8. Patients with implanted pacemaker, defibrillator, nerve stimulator or other active electronic medical devices; sensitive to conductive hydrogels used on electrocardiogram (ECG) stickers or transcutaneous electrical nerve stimulation (TENS) electrodes typically used for TTFields studies.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | from the initiation of study treatment and through study completion, up to 1 year
  evaluate the overall response rate of patients with mUM treated with TTF in combination with nivolumab and ipilimumab.
Overall Safety | From the initiation of study treatment and through study completion, up to 1 year
  Evaluate the safety of TTF in combination with nivolumab and ipilimumab (Number of patients who developed grade 3 treatment-related adverse events as assessed by CTCAE v5)

SECONDARY OUTCOMES:
Overall Survival Rate | From initiation of study treatment until date of death from any cause, up to 100 months
  to assess the median progression free survival and overall survival of treated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Moser, MD, Principal Investigator — HonorHealth Research Institute
Locations (2):
- United States (2):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - The Angeles Clinic and Research Insititute, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No